CLINICAL TRIAL: NCT03916744
Title: A Phase I, Multicenter, Open-Label Preoperative, Short-Term Window Study of GDC-9545 in Postmenopausal Women With Stage I-III Operable, Estrogen Receptor-Positive Breast Cancer
Brief Title: A Study of Giredestrant (GDC-9545) in Postmenopausal Women With Stage I-III Operable, Estrogen Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GO40987; 2018-003798-85 (EudraCT Number)
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Giredestrant 10 mg (Experimental)
  Interventions: Drug: Giredestrant; Procedure: Surgery
- Giredestrant 30 mg (Experimental)
  Interventions: Drug: Giredestrant; Procedure: Surgery
- Giredestrant 100 mg (Experimental)
  Interventions: Drug: Giredestrant; Procedure: Surgery

INTERVENTIONS:
Drug: Giredestrant — Giredestrant will be administered orally once daily (QD) starting on Day 1 up to and including the day of surgery (if allowed per local process) on Day 15 (+/-2 days).
  Other Names: GDC-9545; RO7197597; RG6171
Procedure: Surgery — Breast cancer surgery will take place on Day 15 (+/-2 days).

SUMMARY:
This study will evaluate the pharmacodynamics, pharmacokinetics, safety, and biologic activity of giredestrant in participants with Stage I-III operable estrogen receptor (ER)-positive, human epidermal growth factor receptor 2 (HER2)-negative, untreated breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Histologically confirmed invasive breast carcinoma, with all of the following characteristics: Primary tumor greater than or equal to (≥)1.5 centimeters (cm) in largest diameter by ultrasound; Stage I-III operable breast cancer; Documentation confirming the absence of distant metastasis (M0) as determined by institutional practice.
* ER-positive tumor and HER2-negative breast cancer as per local laboratory testing
* Postmenopausal status
* Breast cancer eligible for primary surgery
* Submission of a representative tumor tissue specimen
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (≤)1
* Adequate organ function

Exclusion Criteria:

* Diagnosis of inflammatory breast cancer
* Diagnosis of bilateral breast cancer
* Concurrent use of hormone replacement therapies
* Previous systemic or local treatment for the primary breast cancer currently under investigation
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study entry
* Current treatment with any systemic anti-cancer therapies
* Major surgery within 4 weeks prior to enrollment
* Radiation therapy within 2 weeks prior to enrollment
* Diagnosis of any secondary malignancy within 3 years prior to enrollment, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or upper gastrointestinal surgery including gastric resection
* Known HIV infection
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* History of allergy to giredestrant or any of its excipients
* Any condition requiring anti-coagulants, such as warfarin, heparin, or thrombolytic drugs
* History of documented hemorrhagic diathesis or coagulopathy
* History or presence of symptomatic bradycardia or sick sinus syndrome
* Baseline heart rate ≤55 beats per minute (bpm) prior to enrollment
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction
* QT interval corrected through use of Fridericia's formula (QTcF) >470 milliseconds demonstrated by at least two ECGs >30 minutes apart
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease, coronary heart disease, clinically significant electrolyte abnormalities, or family history of sudden unexplained death or long QT syndrome
* Current treatment with medications that are well known to prolong the QT interval
* History or presence of uncontrolled hypothyroidism
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (3):
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Sunshine Hospital, St Albans, Victoria
- Belgium (3):
  - Clinique Edith Cavell; Pharmacie, Auderghem
  - UZ Antwerpen, Edegem
  - Clinique Sainte-Elisabeth; Oncologie, Namur
- Spain (5):
  - Onkologikoa - Instituto Oncológico de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional;Servicio de Oncologia, Madrid
  - HM Sanchinarro ? CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Barts Health NHS Trust; William Harvey Heart Centre, QMUL School of Medicine & Dentistry, London
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Giredestrant 10 mg: Giredestrant 10 milligrams (mg) was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
- Giredestrant 30 mg: Giredestrant 30 milligrams (mg) was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
- Giredestrant 100 mg: Giredestrant 100 milligrams (mg) was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
Period: Overall Study
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg
Started (Intent-to-Treat (ITT) Population) | 17 | 40 | 18
Received at Least One Dose of Study Drug (Safety Evaluable Population) | 17 | 40 | 17
Completed | 17 | 39 | 16
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: This is the Intent-to-Treat (ITT) Population, which includes all participants enrolled in the study regardless of whether they received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | Total
Number analyzed (Participants) | 17 | 40 | 18 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age was missing for one participant in the giredestrant 100 mg arm because of early withdrawal from the study.
  Years
    number analyzed (Participants) | 17 | 40 | 17 | 74
    (all) | 63.4 (8.9) | 64.1 (9.4) | 64.1 (7.7) | 63.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 40 | 18 | 75
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 0 | 4
  Not Hispanic or Latino | 4 | 19 | 6 | 29
  Unknown or Not Reported | 13 | 17 | 12 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 16 | 38 | 17 | 71
  Multiple | 1 | 0 | 0 | 1
  Unknown | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline [Count of Participants; unit: Participants] — In order to enroll in the study, a participant was required to have an ECOG performance status ≤1; statuses of 0 and 1 are defined as follows: 0 = Fully active, able to carry on all pre-disease performance without restrictions; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework or office work). Population: ECOG performance status was missing for one participant in the giredestrant 100 mg arm because of early withdrawal from the study.
  Participants
    number analyzed (Participants) | 17 | 40 | 17 | 74
    ECOG Performance Status of 0 | 17 | 36 | 17 | 70
    ECOG Performance Status of 1 | 0 | 4 | 0 | 4
Initial Staging of Breast Cancer (Breast Cancer History) [Count of Participants; unit: Participants] — The TNM description is used to assign an overall stage for breast cancer. There are 5 stages, usually written as Roman numerals: Stage 0 (in-situ breast cancer), followed by Stages I to IV (metastatic breast cancer). Generally, the higher the stage number, the more the cancer has spread. Stage I - the tumor is usually small and hasn't grown outside of the organ it started in. Stages II and III - the tumor is larger or has grown outside of the organ it started in to nearby tissue.
  Participants
    Stage I | 9 | 19 | 10 | 38
    Stage II | 8 | 21 | 7 | 36
    Stage III | 0 | 0 | 1 | 1
Tumor Grade (Breast Cancer History) [Count of Participants; unit: Participants] — The tumor grade is a description of how the cancer cells look compared to normal cells. A pathologist looks at a tissue sample from the tumor under a microscope and assigns a grade ranging from Grade 1 (low) to Grade 3 (high). The higher the grade, the more abnormal the cells look. Higher grade cancer cells tend to grow more quickly and are more likely to spread than low-grade cancer cells.
  Participants
    Grade 1 | 6 | 13 | 4 | 23
    Grade 2 | 9 | 23 | 12 | 44
    Grade 3 | 2 | 4 | 2 | 8
Nodal Status (Breast Cancer History) [Count of Participants; unit: Participants]
  Negative | 14 | 37 | 17 | 68
  Positive | 2 | 3 | 1 | 6
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tumor Cell Proliferation, as Measured by the Proportion of Nuclei Staining Ki67-Positive at Surgery Relative to Baseline in Pre- and Post-Treatment Tumor Biopsy Samples
Description: The biological response to the study treatment was assessed by measuring changes in cell proliferation (Ki67 expression) using formalin-fixed paraffin-embedded histopathology sections of the tumor biopsy specimens taken at baseline and at day of surgery. Baseline was defined as a sample taken prior to initiation of study drug. The results show the proportion of nuclei staining Ki67-positive (Ki67+) in the tumor biopsy sample taken post-treatment (at surgery) relative to that in the pre-treatment sample (at baseline).
Time Frame: Baseline and Surgery (Day 15)
Population: Efficacy Evaluable Population: all participants who 1) had non-missing baseline and post-baseline Ki67 results available, 2) did not discontinue early from the study, 3) had taken at least 12 doses, and 4) had no more than one modified dose. A total of 10 participants (2 in the 10mg cohort, 5 in the 30mg cohort, and 3 in the 100mg cohort) were excluded from efficacy evaluation for not meeting the criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: Proportion of Ki67+ nuclei
Groups:
- All Participants, Efficacy: Giredestrant (10, 30, or 100 mg): This analysis set includes all efficacy-evaluable participants. Participants in the three cohorts received giredestrant (10 mg, 30 mg, or 100 mg) that was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Efficacy: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 15 | 35 | 15 | 65
Proportion of Ki67+ nuclei | 0.20 [0.12 to 0.31] | 0.24 [0.18 to 0.32] | 0.22 [0.13 to 0.37] | 0.22 [0.18 to 0.28]

2. Primary Outcome: Change From Baseline in Tumor Cell Proliferation, as Measured by the Difference in the Percentage of Nuclei Staining Ki67-Positive at Surgery Compared With Baseline in Pre- and Post-Treatment Tumor Biopsy Samples
Description: The biological response to the study treatment was assessed by measuring changes in cell proliferation (Ki67 expression) using formalin-fixed paraffin-embedded histopathology sections of the tumor biopsy specimens taken at baseline and at day of surgery. Baseline was defined as a sample taken prior to initiation of study drug. The results show the percentage of nuclei staining Ki67-positive (Ki67+) in the pre- and post-treatment tumor biopsy samples (taken at baseline and surgery, respectively) and the absolute difference in the percentage of Ki67+ nuclei between the two samples (calculated as surgery minus baseline).
Time Frame: Baseline and Surgery (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of nuclei Ki67+
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Efficacy: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 15 | 35 | 15 | 65
Percentage of nuclei Ki67+
  Baseline (BL) - Value at Visit | 15.70 (9.25) | 15.10 (11.23) | 15.58 (9.95) | 15.35 (10.36)
  Surgery - Value at Visit | 4.22 (4.70) | 4.12 (4.35) | 4.08 (3.80) | 4.13 (4.25)
  Change from BL at Surgery (Surgery minus BL) | -11.49 (7.84) | -10.98 (8.53) | -11.49 (8.23) | -11.21 (8.18)

3. Secondary Outcome: Number of Participants With at Least One Adverse Event and by Severity, Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0)
Description: All adverse events (AEs) were recorded and the investigator independently assessed the seriousness and severity of each AE. AE severity was graded on a scale from 1 to 5 using the NCI-CTCAE v5.0; any events not specifically listed in the scale were defined as: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening; and Grade 5 is death related to an AE. Investigators used their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether an AE was considered to be related to the study drug.
Time Frame: From Baseline to Day 43
Population: Safety Evaluable Population: all participants who received at least one dose of giredestrant. One participant from the ITT population did not receive the study drug because of early withdrawal from the study.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants, Safety: Giredestrant (10, 30, or 100 mg): This analysis set includes all safety-evaluable participants. Participants in the three cohorts received giredestrant (10 mg, 30 mg, or 100 mg) that was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
Participants
  Any Adverse Event (AE) | 12 | 27 | 14 | 53
  AE with Fatal Outcome | 0 | 0 | 0 | 0
  Serious AE | 1 | 2 | 1 | 4
  Related Serious AE | 0 | 0 | 0 | 0
  AE Leading to Withdrawal from Study Drug | 0 | 0 | 0 | 0
  AE Leading to Interruption of Study Drug | 1 | 0 | 1 | 2
  Related AE | 7 | 17 | 8 | 32
  Grade 3-4 AE | 1 | 3 | 1 | 5
  Related Grade 3-4 AE | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Abnormal Vital Signs During Treatment
Description: Vital signs, which included diastolic and systolic blood pressure, pulse rate, and body temperature, were measured while the participant was sitting and according to institutional practices. Any of the vital signs that were outside of the normal reference range (in the specified direction - low or high) were considered abnormalities. Not every abnormality qualified as an adverse event (AE). A vital sign result had to be reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Baseline, Days 1, 8, and 15
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
Percentage of participants
  Diastolic Blood Pressure - Low | 5.9 | 12.5 | 23.5 | 13.5
  Diastolic Blood Pressure - High | 64.7 | 35.0 | 11.8 | 36.5
  Systolic Blood Pressure - High | 82.4 | 70.0 | 58.8 | 70.3
  Pulse Rate - Low | 11.8 | 27.5 | 64.7 | 32.4
  Pulse Rate - High | 0 | 2.5 | 0 | 1.4
  Body Temperature - Low | 88.2 | 82.5 | 94.1 | 86.5

5. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline, Day 8, Surgery (Day 15), and Post-Surgery (Day 43)
Population: Safety Evaluable Population: all participants who received at least one dose of giredestrant. One participant from the ITT population did not receive the study drug because of early withdrawal from the study. The number analyzed indicates all participants who had a non-missing assessment at a given timepoint.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
beats per minute
  Baseline (BL) - Value at Visit | 75.3 (9.5) | 72.6 (11.1) | 72.1 (10.6) | 73.1 (10.6)
  Change from BL at Day 8: number analyzed (Participants) | 16 | 38 | 15 | 69
  Change from BL at Day 8 | 1.4 (8.5) | -1.9 (11.3) | -11.1 (10.6) | -3.1 (11.3)
  Change from BL at Surgery: number analyzed (Participants) | 17 | 37 | 15 | 69
  Change from BL at Surgery | 2.4 (9.7) | -3.8 (10.7) | -13.9 (10.8) | -4.5 (11.8)
  Change from BL at Post-Surgery: number analyzed (Participants) | 17 | 38 | 16 | 71
  Change from BL at Post-Surgery | 2.2 (12.0) | 3.5 (11.4) | 4.2 (11.3) | 3.4 (11.4)
  Change from BL at Post-BL Minimum | -4.2 (9.2) | -7.4 (9.9) | -14.4 (10.7) | -8.3 (10.4)
  Change from BL at Post-BL Maximum | 9.5 (7.2) | 6.7 (11.1) | 4.8 (10.0) | 6.9 (10.1)

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Systolic blood pressure was measured while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline, Day 8, Surgery (Day 15), and Post-Surgery (Day 43)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 135.4 (18.6) | 128.0 (14.2) | 129.4 (14.7) | 130.0 (15.5)
  Change from BL at Day 8: number analyzed (Participants) | 16 | 38 | 15 | 69
  Change from BL at Day 8 | -1.1 (12.3) | 2.9 (14.0) | -7.9 (14.3) | -0.3 (14.2)
  Change from BL at Surgery: number analyzed (Participants) | 17 | 37 | 15 | 69
  Change from BL at Surgery | -2.2 (15.7) | 5.7 (15.2) | -1.4 (17.3) | 2.2 (16.0)
  Change from BL at Post-Surgery: number analyzed (Participants) | 17 | 38 | 16 | 71
  Change from BL at Post-Surgery | -2.1 (14.6) | 1.0 (13.2) | -3.2 (15.3) | -0.7 (13.9)
  Change from BL at Post-BL Minimum | -9.5 (12.0) | -5.5 (11.2) | -12.5 (14.6) | -8.0 (12.4)
  Change from BL at Post-BL Maximum | 5.9 (13.6) | 11.8 (13.4) | 3.2 (15.2) | 8.5 (14.2)

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Diastolic blood pressure was measured while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline, Day 8, Surgery (Day 15), and Post-Surgery (Day 43)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 78.4 (10.3) | 75.2 (10.7) | 76.9 (10.8) | 76.3 (10.6)
  Change from BL at Day 8: number analyzed (Participants) | 16 | 38 | 15 | 69
  Change from BL at Day 8 | -3.4 (7.3) | -0.5 (7.4) | -9.5 (10.3) | -3.1 (8.7)
  Change from BL at Surgery: number analyzed (Participants) | 17 | 37 | 15 | 69
  Change from BL at Surgery | -3.2 (7.9) | -2.1 (12.5) | -8.3 (10.7) | -3.7 (11.2)
  Change from BL at Post-Surgery: number analyzed (Participants) | 17 | 38 | 16 | 71
  Change from BL at Post-Surgery | 4.1 (8.0) | 0.1 (10.5) | -4.5 (9.8) | 0.0 (10.1)
  Change from BL at Post-BL Minimum | -6.4 (6.6) | -6.2 (8.7) | -12.2 (8.5) | -7.6 (8.5)
  Change from BL at Post-BL Maximum | 5.6 (7.0) | 3.8 (10.8) | -2.8 (9.2) | 2.7 (10.1)

8. Secondary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured according to institutional practice. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value. The post-baseline minimum and maximum change from baseline values are, respectively, the smallest and largest value changes obtained after baseline through the last study visit. Baseline was defined as the participant's last value prior to initiation of study drug.
Time Frame: Baseline, Day 8, Surgery (Day 15), and Post-Surgery (Day 43)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: degrees Celsius (C)
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
degrees Celsius (C)
  Baseline (BL) - Value at Visit | 36.36 (0.48) | 36.41 (0.38) | 36.25 (0.24) | 36.36 (0.38)
  Change from BL at Day 8: number analyzed (Participants) | 16 | 38 | 15 | 69
  Change from BL at Day 8 | -0.03 (0.41) | -0.06 (0.51) | -0.09 (0.43) | -0.06 (0.47)
  Change from BL at Surgery: number analyzed (Participants) | 17 | 37 | 15 | 69
  Change from BL at Surgery | 0.14 (0.51) | -0.09 (0.46) | -0.18 (0.43) | -0.05 (0.47)
  Change from BL at Post-Surgery: number analyzed (Participants) | 17 | 38 | 16 | 71
  Change from BL at Post-Surgery | -0.03 (0.56) | -0.05 (0.39) | -0.11 (0.50) | -0.06 (0.45)
  Change from BL at Post-BL Minimum | -0.20 (0.52) | -0.34 (0.44) | -0.39 (0.42) | -0.32 (0.45)
  Change from BL at Post-BL Maximum | 0.28 (0.42) | 0.15 (0.44) | 0.12 (0.32) | 0.17 (0.41)

9. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities in Hematology Tests During Treatment, Among Participants Without the Abnormality at Baseline
Description: Laboratory parameters for hematology will be measured and compared with a standard reference range. Any of the laboratory test results that were outside of a parameter's normal reference range (in the specified direction - low or high) were considered abnormalities. Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Baseline, Days 1, 8, and 15
Population: Safety Evaluable Population: the number of participants analyzed includes all participants who received at least one dose of giredestrant. The number analyzed for a given laboratory parameter represents the number of participants without an abnormality (in the specified direction) at baseline for that parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
Percentage of participants
  Hematocrit - Low: number analyzed (Participants) | 10 | 31 | 8 | 49
  Hematocrit - Low | 0 | 3.2 | 0 | 2.0
  Hematocrit - High: number analyzed (Participants) | 9 | 31 | 7 | 47
  Hematocrit - High | 22.2 | 0 | 0 | 4.3
  Hemoglobin - Low: number analyzed (Participants) | 10 | 31 | 8 | 49
  Hemoglobin - Low | 10.0 | 0 | 0 | 2.0
  Hemoglobin - High: number analyzed (Participants) | 9 | 32 | 8 | 49
  Hemoglobin - High | 0 | 3.1 | 0 | 2.0
  Lymphocytes, Absolute Count (Abs) - Low: number analyzed (Participants) | 10 | 32 | 8 | 50
  Lymphocytes, Absolute Count (Abs) - Low | 0 | 3.1 | 0 | 2.0
  Lymphocytes, Abs - High: number analyzed (Participants) | 10 | 31 | 8 | 49
  Lymphocytes, Abs - High | 0 | 3.2 | 12.5 | 4.1
  Neutrophils, Total, Abs - Low: number analyzed (Participants) | 10 | 31 | 8 | 49
  Neutrophils, Total, Abs - Low | 0 | 3.2 | 0 | 2.0
  Erythrocytes - Low: number analyzed (Participants) | 9 | 30 | 8 | 47
  Erythrocytes - Low | 22.2 | 6.7 | 0 | 8.5
  Total Leukocyte Count - Low: number analyzed (Participants) | 10 | 32 | 8 | 50
  Total Leukocyte Count - Low | 0 | 3.1 | 0 | 2.0

10. Secondary Outcome: Percentage of Participants With Laboratory Abnormalities in Blood Chemistry and Coagulation Tests During Treatment, Among Participants Without the Abnormality at Baseline
Description: Laboratory parameters for blood chemistry and coagulation were measured and compared with a standard reference range. Any of the laboratory test results that were outside of a parameter's normal reference range (in the specified direction - low or high) were considered abnormalities. Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. SGPT/ALT = alanine aminotransferase; SGOT/AST = aspartate aminotransferase
Time Frame: Baseline, Days 1, 8, and 15
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 17 | 40 | 17 | 74
Percentage of participants
  Albumin - Low: number analyzed (Participants) | 10 | 30 | 8 | 48
  Albumin - Low | 0 | 3.3 | 0 | 2.1
  Albumin - High: number analyzed (Participants) | 10 | 30 | 8 | 48
  Albumin - High | 0 | 3.3 | 0 | 2.1
  Alkaline Phosphatase - High: number analyzed (Participants) | 8 | 29 | 6 | 43
  Alkaline Phosphatase - High | 0 | 3.4 | 0 | 2.3
  SGPT/ALT - High: number analyzed (Participants) | 9 | 30 | 7 | 46
  SGPT/ALT - High | 0 | 6.7 | 14.3 | 6.5
  SGOT/AST - High: number analyzed (Participants) | 9 | 32 | 7 | 48
  SGOT/AST - High | 0 | 3.1 | 14.3 | 4.2
  Bicarbonate HCO3 - Low: number analyzed (Participants) | 9 | 32 | 8 | 49
  Bicarbonate HCO3 - Low | 0 | 3.1 | 0 | 2.0
  Bicarbonate HCO3 - High: number analyzed (Participants) | 6 | 21 | 5 | 32
  Bicarbonate HCO3 - High | 16.7 | 9.5 | 40.0 | 15.6
  Blood Urea Nitrogen - High: number analyzed (Participants) | 10 | 32 | 7 | 49
  Blood Urea Nitrogen - High | 10.0 | 3.1 | 0 | 4.1
  Calcium - High: number analyzed (Participants) | 9 | 32 | 8 | 49
  Calcium - High | 0 | 3.1 | 0 | 2.0
  Carbon Dioxide - High: number analyzed (Participants) | 3 | 4 | 1 | 8
  Carbon Dioxide - High | 33.3 | 25.0 | 0 | 25.0
  Chloride - Low: number analyzed (Participants) | 10 | 31 | 8 | 49
  Chloride - Low | 10.0 | 3.2 | 12.5 | 6.1
  Chloride - High: number analyzed (Participants) | 8 | 32 | 8 | 48
  Chloride - High | 0 | 9.4 | 0 | 6.3
  Creatinine - High: number analyzed (Participants) | 10 | 32 | 8 | 50
  Creatinine - High | 0 | 3.1 | 0 | 2.0
  Direct Bilirubin - Low: number analyzed (Participants) | 10 | 26 | 6 | 42
  Direct Bilirubin - Low | 10.0 | 0 | 0 | 2.4
  Direct Bilirubin - High: number analyzed (Participants) | 9 | 29 | 8 | 46
  Direct Bilirubin - High | 11.1 | 3.4 | 0 | 4.3
  Glucose, Fasting - High: number analyzed (Participants) | 6 | 16 | 4 | 26
  Glucose, Fasting - High | 0 | 31.3 | 0 | 19.2
  Glucose, Fasting Unknown - High: number analyzed (Participants) | 3 | 14 | 3 | 20
  Glucose, Fasting Unknown - High | 33.3 | 21.4 | 33.3 | 25.0
  Magnesium - High: number analyzed (Participants) | 10 | 32 | 8 | 50
  Magnesium - High | 0 | 0 | 12.5 | 2.0
  Phosphorus - Low: number analyzed (Participants) | 10 | 32 | 8 | 50
  Phosphorus - Low | 10.0 | 0 | 0 | 2.0
  Phosphorus - High: number analyzed (Participants) | 10 | 31 | 8 | 49
  Phosphorus - High | 0 | 3.2 | 0 | 2.0
  Potassium - High: number analyzed (Participants) | 10 | 32 | 8 | 50
  Potassium - High | 0 | 3.1 | 0 | 2.0
  Sodium - Low: number analyzed (Participants) | 10 | 32 | 8 | 50
  Sodium - Low | 0 | 3.1 | 0 | 2.0
  Bilirubin - High: number analyzed (Participants) | 10 | 30 | 8 | 48
  Bilirubin - High | 0 | 6.7 | 0 | 4.2
  Protein, Total - Low: number analyzed (Participants) | 8 | 30 | 7 | 45
  Protein, Total - Low | 0 | 3.3 | 0 | 2.2
  Protein, Total - High: number analyzed (Participants) | 10 | 31 | 8 | 49
  Protein, Total - High | 0 | 3.2 | 0 | 2.0
  Prothrombin Time - High: number analyzed (Participants) | 17 | 33 | 14 | 64
  Prothrombin Time - High | 0 | 3.0 | 0 | 1.6
  International Normalized Ratio - High: number analyzed (Participants) | 17 | 39 | 15 | 71
  International Normalized Ratio - High | 0 | 2.6 | 0 | 1.4
  Activated Partial Thromboplastin Time - Low: number analyzed (Participants) | 15 | 37 | 17 | 69
  Activated Partial Thromboplastin Time - Low | 13.3 | 16.2 | 11.8 | 14.5

11. Secondary Outcome: Percentage of Participants With Abnormal Electrocardiogram Parameters During Treatment
Description: Electrocardiogram (ECG) recordings were performed after the participant had been resting in a supine position for at least 10 minutes. ECG parameters included heart rate, PR and QRS durations, and QT and QTcF intervals. Per the protocol, ECG readings post-treatment were limited to those for whom it was clinically indicated. Any of the ECG parameters that were outside of the normal reference range (in the specified direction - low or high) were considered abnormalities. Not every abnormality qualified as an adverse event (AE). An ECG test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment.
Time Frame: Baseline, Days 1, 8, and 15
Population: The analysis included a small number of participants who had ECG readings post-treatment because, per the protocol, ECGs were limited to those for whom it was clinically indicated.
Measure: Number; unit: Percentage of participants
Groups:
- All Participants, Safety (ECG): Giredestrant (10, 30, or 100 mg): This analysis set includes a subset of the safety-evaluable participants who had electrocardiogram (ECG) readings post-treatment because, per the protocol, ECGs were limited to those for whom it was clinically indicated. Participants in the three cohorts received giredestrant (10 mg, 30 mg, or 100 mg) that was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety (ECG): Giredestrant (10, 30, or 100 mg)
Number analyzed (Participants) | 8 | 7 | 4 | 19
Percentage of participants
  PR Duration - Low | 12.5 | 0 | 0 | 5.3
  PR Duration - High | 0 | 0 | 25.0 | 5.3

12. Secondary Outcome: Plasma Concentration of Giredestrant at Steady State by Dose Level
Description: Plasma samples were obtained on the day of surgery (Day 15), or prior to biopsy on Day 14.
Time Frame: Predose on day of surgery (Day 15), or prior to biopsy (Day 14)
Population: The Pharmacokinetics Analysis Population consisted of all participants who received at least one dose of giredestrant and had a measurable concentration at the specific timepoint collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg
Number analyzed (Participants) | 16 | 36 | 17
nanograms per millilitre (ng/mL) | 58.8 (58.1) | 130 (59.1) | 441 (71.2)

ADVERSE EVENTS:
Time Frame: From Baseline to Day 43
Groups:
- All Participants, Safety: Giredestrant (10, 30, or 100 mg): This analysis set includes a subset of the safety-evaluable participants who had ECG readings post-treatment because, per the protocol, ECGs were limited to those for whom it was clinically indicated. Participants in the three cohorts received giredestrant (10 mg, 30 mg, or 100 mg) that was administered orally once daily up to and including the day of surgery (if allowed per local process) on Day 15. Surgery should have been performed within 24 hours after the last dose of giredestrant. Following surgery, participants had a post-surgery follow-up visit after a period of 28 days.
Arm/Group | Giredestrant 10 mg | Giredestrant 30 mg | Giredestrant 100 mg | All Participants, Safety: Giredestrant (10, 30, or 100 mg)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/40 | 0/17 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/40 | 1/17 | 4/74
Other Adverse Events (participants affected / at risk) | 12/17 | 21/40 | 14/17 | 47/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant 10 mg (N=17) | Giredestrant 30 mg (N=40) | Giredestrant 100 mg (N=17) | All Participants, Safety: Giredestrant (10, 30, or 100 mg) (N=74)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant 10 mg (N=17) | Giredestrant 30 mg (N=40) | Giredestrant 100 mg (N=17) | All Participants, Safety: Giredestrant (10, 30, or 100 mg) (N=74)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1) | 9 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 5 (5) | 8 (8)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3) | 6 (6)
Product dose omission in error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Breast discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03916744/Prot_SAP_000.pdf